CLINICAL TRIAL: NCT05451316
Title: A Study to Evaluate Effectiveness of Upadacitinib in Moderate to Severe AD With Prurigo Nodularis in the Real World in Japan
Brief Title: A Study to Assess Change in Disease Activity in Adolescents and Adults With Moderate to Severe Prurigo-type Atopic Dermatitis in Japan Who Are Treated With Oral Upadacitinib
Acronym: ADMIRE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-433
Record Dates: First submitted 2022-07-07; First posted 2022-07-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Prurigo Nodularis; Prurigo-type AD; Skin; Dermatology; Upadacitinib; ADMIRE; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Upadacitinib: Adolescents and adults with moderate to severe prurigo-type AD, who are prescribed UPA according to the label and practice in Japan.

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Around one-third of patients with AD have had at least 1 incidence of prurigo nodularis (PN), which is characterized by intense, persistent itchy skin and sometimes pain with burning. In this study, the effectiveness of upadacitinib (UPA) will be assessed in participants with prurigo-type AD in a real world (RW) setting in Japan.

UPA is an approved drug for the treatment of AD. Adults and adolescents who have been diagnosed with prurigo-type AD and prescribed UPA according to the label and practice in Japan will be enrolled in this observational study. The doctor's decision to prescribe UPA will be made prior to and independently of study participation. Approximately 200 participants will be enrolled in the study at 10 sites in Japan.

Participants will receive extended-release oral tablets of UPA once-daily for 48 weeks.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed diagnosis of moderate to severe atopic dermatitis (AD) at baseline
* AD symptom onset > 1 year prior to baseline
* Initiation of UPA treatment for AD is indicated and prescribed per the label in Japan
* Worst Pruritus Numerical Rating Scale (WP-NRS) ≥ 4 at baseline
* Presence of palpable prurigo nodules at baseline

Exclusion Criteria:

* Prior treatment with UPA
* Contraindications to UPA
* Chronic pruritus resulting from another condition (e.g., neuropathic disorders) than AD, prurigo nodularis (PN)
* PN caused by medication, metal allergy, infection, insect bite
* Current participation in interventional research

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and adults, age ≥ 12 years, with a physician-confirmed diagnosis of atopic dermatitis (AD), who are prescribed UPA according to the label and practice in Japan. The decision to prescribe UPA will be made prior to and independent of study participation
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving Worst Pruritus Numerical Rating Scale (WP-NRS) reduction ≥ 4. | Up to Week 12
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours in patients with moderate to severe AD, based on the following question: "On a scale 0 to 10, with 0 being 'no itch' and 10 being 'worst imaginable itch', how would you rate your itch at its worst during the past 24 hours?"

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Tohoku Medical and Pharmaceuti /ID# 252486, Sendai, Miyagi, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/